CLINICAL TRIAL: NCT00458510
Title: An Open-Label Study Investigating Long-Term Safety and Tolerability of Fentanyl Citrate Nasal Spray in the Treatment of BTCP in Subjects Taking Regular Opioid Therapy
Brief Title: Long Term Safety Study of Nasalfent (Fentanyl Citrate Nasal Spray) for Treatment of Breakthrough Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Archimedes Development Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CPO45/06/FCNS
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Cancers, Pain
Keywords: Pain; Cancer; Breakthrough
MeSH Terms: conditions — Neoplasms; Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fentanyl, Open-Label treatment (Experimental): All patients take NasalFent at effective dose to treat up to four episodes of breakthrough cancer pain per day
  Interventions: Drug: Fentanyl (Nasalfent, Fentanyl Citrate Nasal Spray)

INTERVENTIONS:
Drug: Fentanyl (Nasalfent, Fentanyl Citrate Nasal Spray) — treatment of up to 4 episodes of pain per day
  Other Names: FCNS

SUMMARY:
Cancer patients taking regular medication for their pain often still have episodes of severe pain that 'break through' despite their background pain treatment. Fentanyl is a strong, short-acting pain killer often used to treat this 'breakthrough' pain. Nasalfent contains fentanyl in a patented drug delivery system called PecSys and is given via a simple nasal spray. This study will examine the long-term safety of Nasalfent in the treatment of breakthrough cancer pain.

DETAILED DESCRIPTION:
Current treatments for breakthrough cancer pain (BTCP) work too slowly to meet the fast onset of most BTCP episodes, they continue to act longer than the episode of pain lasts and so can have unwanted side effects due to this 'over treatment' of the pain episode. In addition most cancer patients have oral problems which make taking pain relief medication by mouth uncomfortable for the patient. Nasalfent is administered via the nose as a simple spray and can be taken by patients or given by their carers. The nasal route is a common way to administer medication for example in the treatment of migraine or allergy. At any time during the study the patient may take their regular treatment for BTCP should they so wish.

This study will examine the long-term safety of Nasalfent treatment for breakthrough cancer pain.

After the study is completed, patients may continue to take medication if their doctor feels it is in the patient's best interest to do so. Safety information will continue to be collected during this period. Treatment may continue on study for as long as the patient requires treatment or until Nasalfent becomes commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give consent
* Women of childbearing potential must have a) negative urine pregnancy test b) not be breast feeding c) agree to practice a reliable form of contraception
* Diagnosis of cancer
* Taking at least 60mg oral morphine or equivalent as 24 hour treatment for cancer-related pain
* Experiencing on average 1 - 4 episodes of breakthrough cancer pain per day usually controlled by rescue pain medication
* Able (or via caregiver) to evaluate and record pain relief, assess medication performance at set times after dosing, record adverse events, record each use of the study drug or rescue medication in a diary
* Able to be up and about for 50% of the day or greater

Exclusion Criteria:

* Intolerance to opioids or fentanyl
* rapidly increasing/uncontrolled pain
* pain that is not cancer related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2007-01; Primary Completion 2011-10 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Long term Safety, tolerability and acceptability | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Russell K Portenoy, MD, Principal Investigator — Beth Israel Medical Center, New York, United States

REFERENCES:
- [Result] Taylor D, Radbruch L, Revnic J, Torres LM, Ellershaw JE, Perelman MS. Long-term use of fentanyl pectin nasal spray in patients with breakthrough pain in cancer [abstract]. J Clin Oncol. 2013:31(15 Suppl);9563